CLINICAL TRIAL: NCT00172016
Title: A Study to Evaluate the Efficacy and Tolerability of Zoledronic Acid in Patients With Metastatic Prostate Cancer Who Can be Treated With a Group of Medications Known as Bisphosphonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EHU01
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer With at Least One Bone Lesion in Patients Receiving Hormonal Therapy and Treatment With Bisphosphonates is Indicated
Keywords: Zoledronic acid; SRE; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- ZOL446 (zoledronic acid) (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
The purpose of this study is to assess the efficacy and tolerability of zoledronic acid in preventing skeletal-related events in patients with prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained
* Age > 18 years
* Histologically confirmed diagnosis of carcinoma of the prostate
* Current (or previous) objective evidence of metastatic disease to the bone
* Currently receiving 1st line hormonal therapy with LHRH agonists or other hormonal treatments
* ECOG performance status of 0, 1, or 2

Exclusion Criteria:

* Patients with abnormal renal function as evidenced by either a serum creatinine determination 1.5 x or greater above the upper limit of normal or by a calculated creatinine clearance of 60 ml/minute or less
* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L)
* WBC<3.0x1'000'000'000, ANC < 1500/mm3, Hgb<8.0 g/dL, platelets < 75 x 1'000'000'000/L.
* Liver function tests >2.5 ULN, serum creatinine >1.5 ULN.
* Patients with another nonmalignant disease which would confound the evaluation of primary endpoints or prevent the patient complying with the protocol.
* Known hypersensitivity to zoledronic acid or other bisphosphonates
* Subjects who, in the opinion of the investigator, are unlikely to cooperate fully during the study

Other protocol-defined inclusion / exclusion criteria apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-01; Primary Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals